CLINICAL TRIAL: NCT01164904
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Ascending Single Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 181 in Healthy Subjects and Subjects With Mild to Moderate Ulcerative Colitis
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 181 in Healthy Subjects and Subjects With Mild to Moderate Ulcerative Colitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 20090107
Record Dates: First submitted 2010-07-01; First posted 2010-07-19 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Ulcerative Colitis
Keywords: Inflammatory Bowel Disease; Amgen
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — abrilumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Experimental (Experimental): Ten escalating dose levels of AMG 181 administered as a single dose SC or IV in healthy volunteers and SC in subjects with mild-to-moderate ulcerative colitis.
  Interventions: Drug: Amg 181

INTERVENTIONS:
Drug: Amg 181 — Ten escalating dose levels of AMG 181 administered as single dose SC or IV, in healthy volunteers and SC subjects with mild-to-moderate ulcerative colitis.

SUMMARY:
To assess the safety and tolerability of single subcutaneous (SC) and intravenous (IV) doses of AMG 181 in healthy subjects and of a single SC dose in subjects with mild to moderate ulcerative colitis (UC)

ELIGIBILITY:
Inclusion Criteria: Healthy Volunteers

* Healthy male or female subjects of non-reproductive potential between 18 to 45 year-of -age
* Body Mass Index (BMI) between 18 and 34 kg/m2
* Normal physical and neurological examination, clinical laboratory values and ECG
* Additional inclusion criteria apply

Inclusion Criteria: Subjects with Mild to Moderate Ulcerative Colitis

* Male or female subjects between 18 to 55 year-of -age
* Body Mass Index (BMI) between 18 and 34 kg/m2
* Diagnosis of Ulcerative Colitis for at least 2 months
* Active, mild to moderate disease as defined by an Ulcerative Colitis Disease Activity Index (UCDAI, aka Mayo score) score of 4 to 9 (inclusive), with a minimum sigmoidoscopy score of 1
* Additional inclusion criteria apply

Exclusion criteria: Healthy Volunteers

* History or evidence of a clinically significant disorder (including psychiatric), condition or disease that would pose a risk to subject safety or interfere with the study evaluations, procedures or completion
* History of malignancy of any type, other than in situ cervical cancer or surgically excised non-melanomatous skin cancers within the past 5 years
* Recent or on-going infection(s)
* Underlying condition(s) that predisposes the subject to infections
* Additional exclusion criteria apply

Exclusion criteria: Subjects with Mild to Moderate Ulcerative Colitis

* Disease limited to the rectum, i.e. within 20 cm of the anal verge
* Any prior gastrointestinal surgery
* Evidence of severe disease (as evidenced by an Hb concentration <11g/dL; toxic megacolon, or an UCDAI score≥10)
* Immunosuppressive therapy with either azathioprine, methotrexate, or mercaptopurine, within the past 3 months
* Prior exposure to a biologic agent or cyclosporine A
* Use of antibiotics within the past 2 weeks of screening and during screening period
* Use of topical (e.g. suppository or enema) mesalamine or steroids within two weeks prior to day 1
* Additional exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2010-07; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of single subcutaneous (SC) and intravenous (IV) doses of AMG 181 in healthy subjects and of a single SC dose in subjects with mild to moderate ulcerative colitis (UC) | Through study completion

SECONDARY OUTCOMES:
To characterize the pharmacokinetics (PK) of ascending single doses of AMG 181 | Through study completion
To characterize the pharmacodynamic (PD) effects of AMG 181 on receptor occupancy and on cell counts in selected lymphocyte subset populations | Through study completion

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (10):
- United States (4):
  - Research Site, Glendale, California
  - Research Site, Danbury, Connecticut
  - Research Site, Plymouth, Minnesota
  - Research Site, Duncansville, Pennsylvania
- Australia (4):
  - Research Site, Herston, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Prahran, Victoria
  - Research Site, Nedlands, Western Australia
- New Zealand (2):
  - Research Site, Auckland
  - Research Site, Christchurch

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com